CLINICAL TRIAL: NCT07323160
Title: Determining the Effect of Discharge Education Provided Using the Teaching-back Method on Readmission Rates and Patient Satisfaction in Patients Undergoing Same-day Anal Fistula Surgery
Brief Title: Determining the Effect of Education Given to Patients Undergoing Outpatient Anal Fistula Surgery
Acronym: anal fistula
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Cemile Yaşar, surgical Nurse, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MSKU Ethics Committe No:250098
Record Dates: First submitted 2025-11-14; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Anal Fistula; Patient Discharge Education; Outpatient Anal Surgery
Keywords: Anal fistula, Day surgery, Discharge teaching, Patient satisfaction, Readmission
MeSH Terms: conditions — Rectal Fistula; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Two parallel groups: teach-back discharge education vs. routine discharge education.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach-back discharge education (Experimental): Participants receive discharge education using the teach-back method.
  Interventions: Behavioral: Teach-back discharge education
- Routine discharge education (No Intervention): Participants receive routine discharge education.

INTERVENTIONS:
Behavioral: Teach-back discharge education — For the Experimental Group:
  Intervention Name: Teach-back discharge education
  Intervention Type: Behavioral
  Description: Discharge education provided using the teach-back method.
  For the Control Group:
  Intervention Name: Routine discharge education
  Intervention Type: Behavioral
  Description: Standard discharge education provided without teach-back.
  Arms: Teach-back discharge education

SUMMARY:
It is emphasized that discharge education should shift from traditional healthcare provider-centered, one-way education to patient-centered education based on patient-care provider interaction to ensure patients' active participation in their own care, adherence to the recommended treatment plan, and maintenance of surgical success after outpatient anal fistula surgery. In this context, it is suggested that an effective education method such as teach-back can be used in clinical settings to teach patients complex health information and facilitate their understanding of discharge education. While studies exist in the literature evaluating the impact of health literacy after general surgery, no studies have been found specifically evaluating health literacy and discharge education for anal fistula surgery. Furthermore, it is emphasized that further research is needed to improve the quality of postoperative care after anal fistula surgery and to better understand the factors contributing to unplanned hospital returns. Based on this need, this study is a randomized controlled trial with a pretest and posttest approach aimed at determining the effect of teach-back-based discharge education on hospital readmission and patient satisfaction in outpatient anal fistula surgery patients. The study sample was calculated as a total of 68 people, 34 in each group, based on a power analysis performed with the GPower 3.1. 9.7 program, using a type 1 error of 0.05, a type 2 error of 0.20, and an effect size of 0.70 to determine the difference in measurements between the groups. Considering the possible attrition in the study, the sample size was increased by 10%, and a total of 76 people, 38 in each group, were planned to be included in the study. Following Ethics Committee approval and institutional permissions, the study data will be collected using the Individual Identification Form, Health Literacy Scale, Anal Fistula Surgery Discharge Education Knowledge Test, Discharge Satisfaction Scale, and Post-Discharge Follow-up Form, from patients scheduled for and undergoing outpatient anal fistula surgery at Muğla Training and Research Hospital between November 15, 2025, and January 30, 2027. The research will be conducted in three phases: the development of the education brochure and knowledge test, and the preoperative and postoperative phases. The "Anal Fistula Surgery Discharge Education Knowledge Test" was developed to assess patients' knowledge of anal fistula and its care. The "Anal Fistula Surgery Discharge Education Patient Booklet" was developed by the researchers using literature review and consultation with a General Surgery Specialist specializing in anal fistulas to provide specific training on anal fistula surgery and postoperative care. These were then sent to specialists for expert opinion. All patients presenting to the General Surgery Outpatient Clinic for anal fistula surgery who meet the inclusion criteria will be interviewed face-to-face before surgery to be informed about the study. Patients who agree to participate will be asked to sign a consent form. Because outpatient surgeries involve admission and discharge within 24 hours, and patients arrive at the Proctology Unit on the day of surgery, all patients will be summoned to the General Surgery Outpatient Clinic the day before surgery and will complete the "Individual Identification Form," "Health Literacy Scale," and "Anal Fistula Surgery Discharge Education Knowledge Test." Patients will be assigned to the intervention (discharge education via teach-back) and control groups using a block randomization table based on their order of admission to the Proctology Unit for the surgical procedure. Patients in the intervention group will receive discharge education via teach-back using the "Anal Fistula Surgery Discharge Education Patient Booklet." Education will continue until the patient accurately recounts the information to the principal investigator and is confident that the patient has understood the instruction correctly. The control group will receive standard patient education in the clinic and will not receive any intervention. Postoperatively, all patients in both groups will complete the "Anal Fistula Surgery Discharge Education Knowledge Test" post-test and the Discharge Education Satisfaction Scale before being discharged from the unit. Patients in both groups will be contacted weekly for 30 days to monitor their progress. Because the study will provide training, blinding of the assessments will not be possible.

DETAILED DESCRIPTION:
Day surgery refers to surgical procedures in which the patient is admitted to the clinic on the same day, undergoes surgery, and is discharged within 24 hours. This approach is increasingly being implemented due to its cost-effectiveness, reduced risk of infection, minimally invasive nature, faster recovery, lower risk, and shorter hospital stay. One type of surgery currently performed on a day case basis is anorectal surgery, including anal fistula surgery.

An anal fistula is characterized by a chronic infection between the anorectal canal and the perianal skin. It often develops after a perianal abscess and carries a high risk of recurrence. Complex anal fistulas, due to their anatomical complexity, pose significant complications and risks not only from a surgical perspective but also from a nursing care perspective. These patients require careful management due to high recurrence rates, post-treatment complications, and decreased quality of life. Studies on the subject indicate that anal fistula patients experience chronic complaints such as pain, discharge, recurrence, and a decrease in quality of life. These complaints can lead to social isolation, depression, and sleep disturbances. The disrupted sleep patterns and limitations in daily activities caused by pain and drainage significantly impact these patients' quality of life. Therefore, the importance of providing individualized education, such as supporting patients with educational brochures and providing emergency contact information, is emphasized to ensure active participation in their own care after anal fistula surgery, adherence to the recommended treatment plan, and maintenance of surgical success. Furthermore, while outpatient surgeries reduce hospital costs and increase patient satisfaction, they also reduce the time healthcare professionals spend with the patient. This limits patient interaction with healthcare professionals and leads to increased caregiving responsibilities being assigned to the patient and their families. During this period, patients' lack of knowledge and inadequate education regarding the post-discharge period leads to postoperative pain, bleeding, wound care, medication management, anal hygiene, and difficulty recognizing signs of complications, leading to re-admissions to the hospital, increased risk of complications, and prolonged recovery. Patient education, a crucial aspect of clinical practice and patient care, is crucial for ensuring continuity of care for these patients, supporting their recovery at home, and preventing the risk of recurrence, complications, and hospital readmissions. This highlights the importance of nurses involved in the care of these patients to take an active role not only in physical care practices but also in patient education, psychosocial support, and postoperative follow-up. Despite education on care and complications after anal fistula surgery, patients are reported to experience anxiety regarding issues such as bleeding, pain, and wound care and tend to forget 40-80% of the information provided. Furthermore, existing studies indicate that education generally focuses on surgical technique and anatomical factors, while factors directly related to nursing care and education, such as patient education and health literacy, are not adequately addressed. Health education is an intervention that empowers individuals to actively participate in decision-making processes regarding their own health and is a fundamental element of nursing care. Discharge education, a key component of health education, increases patient awareness of potential postoperative complications and their early symptoms, supports self-care at home, and accelerates the recovery process. It also contributes to improving health outcomes, including hospital readmissions, and enhancing patient satisfaction. To achieve this, it is emphasized that discharge education should shift from traditional healthcare provider-centered, one-way education to patient-centered education based on patient-caregiver interaction. Therefore, the Agency for Healthcare Research and Quality recommends using an effective education method, such as the teach-back method, to teach patients complex health information in clinical settings and facilitate their understanding of discharge education. Teach-back is a patient-centered education strategy used to teach patients complex health information. This method allows healthcare providers to confirm whether they are educating the patient correctly and how accurately the patient understands the health information. Furthermore, consistently re-educating patients about misunderstood information helps them better remember information. Education using this method has been associated with positive health outcomes, including self-care and the use of healthcare resources. However, for patient education to be effective, the level of health literacy, which defines an individual's capacity to understand, interpret, evaluate, and apply health information and directly impacts their adherence to treatment, should also be considered. Studies indicate that individuals with inadequate health literacy levels struggle to understand and implement recommendations for post-discharge care. They struggle to perform tasks such as understanding physician instructions, reading patient information leaflets, and following post-operative care procedures. This leads to complications, re-admissions, and increased costs. While studies evaluating the impact of health literacy after general surgery exist, no studies specifically evaluating health literacy and discharge education for anal fistula surgery are available. Furthermore, further research is needed to improve the quality of postoperative care after anal fistula surgery and to better understand the factors contributing to unplanned hospital returns. This randomized controlled study, designed to address this need, aimed to determine the impact of discharge education provided through the teach-back method on hospital re-admissions and patient satisfaction in outpatient anal fistula surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Having a day surgery planned, Being admitted to the Proctology Unit for anal fistula surgery, Being undergoing elective anal fistula surgery for the first time, Being planned to have a surgical procedure performed with local anesthesia, Being over 18 years of age, Being able to read and understand Turkish, Being able to read and understand the research instructions, Being literate, Agreeing to participate in the research.

Exclusion Criteria:

* Having surgery planned with general anesthesia, Requiring general anesthesia during the surgical procedure, Being hospitalized for more than 24 hours, Having a recurrent anal fistula, Having another anorectal disease besides the anal fistula, such as advanced Crohn's disease or colorectal cancer, Having complications within 24 hours of surgery and rescheduling surgery, Having visual, auditory, or cognitive problems, Having agreed to participate in the study but wishing to withdraw during follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Effect of teach-back discharge education on postoperative readmission and patient satisfaction | Within 30 days after surgery
  The rate of hospital readmissions within the follow-up period and the mean patient satisfaction scores will be compared between the teach-back discharge education group and the routine discharge education group to evaluate the effect of the intervention.
Discharge Education Satisfaction Scale | within 30 days after surgery
  Discharge Education Satisfaction Scale (TEMÖ): It was developed by Meşe and Köşgeroğlu in 2018 to determine the satisfaction of patients or their relatives who underwent surgical intervention with discharge education. The scale items include 21 items related to the discharge process, home care, medication, pain, infection, exercise, and postoperative follow-up. The minimum score that can be obtained from the scale is 21, and the maximum score is 105. TEMÖ is a 5-point Likert-type scale, and the scale items are scored as "completely satisfied" (5), "satisfied" (4), "partially satisfied" (3), "not satisfied" (2), and "not satisfied at all" (1). The scale has no cut-off point, and higher scores indicate higher satisfaction with discharge education. The Cronbach's alpha coefficient was 0.91 in the original scale, and total item correlation scores were found to range between 0.42 and 0.64 (Meşe, 2018). Permission was obtained from Sevinç Meşe for the use of the scale in the study.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a small sample and includes identifiable information that cannot be fully anonymized. Only summary results will be available.